CLINICAL TRIAL: NCT05361798
Title: A Phase II Study Evaluating T-Cell Clonality After Stereotactic Body Radiation Therapy Alone and in Combination With the Immunocytokine M9241 in Localized High and Intermediate Risk Prostate Cancer Treated With Androgen Deprivation Therapy
Brief Title: T-Cell Clonality After Stereotactic Body Radiation Therapy Alone and in Combination With the Immunocytokine M9241 in Localized High- and Intermediate-Risk Prostate Cancer Treated With Androgen Deprivation Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000114; 000114-C
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Cancer Of Prostate
Keywords: Immunotherapy + Radiation; Combination Therapy; Cancer Of Prostate; Nhs-Il 12
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Arm 1 (Experimental): De-escalating doses of M9241 if appropriate + SBRT
  Interventions: Drug: M9241; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- 2/Arm 2a (Experimental): Highest tolerated dose of M941+SBRT
  Interventions: Drug: M9241; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- 3/Arm 2b (Experimental): SBRT
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: M9241 — In the safety lead in, M9241 will be given in de-escalating doses (starting dose 16.8 mcg/kg, and de-escalated if needed to 12 mcg/kg, or 8 mcg/kg) every 4 weeks for 3 doses. Within 4 weeks after completing SBRT, those participants receiving immunotherapy agents will receive M9241 by subcutaneous injection at dose determined during the safety lead in every 4 weeks for 3 doses.
  Arms: 1/Arm 1; 2/Arm 2a
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT to the prostate will be delivered in 5 fractions of radiation each of 7.25-8.0 Gy, every other day over the course of 10 business days (2-3 weeks). The total dose will be 36.25-40 Gy

SUMMARY:
Background:

Prostate cancer is often treated with radiation and ADT (ADT is androgen deprivation therapy). Up to 30% of these cancers recur within 5 years of treatment. Researchers want to see if a new drug (M9241) can help the immune system to fight prostate cancer.

Objective:

To find what doses of M9241 are safe in people who are treated for prostate cancer. Also, to see what effects M9241 has on the immune system.

Eligibility:

People aged 18 and older with high- and intermediate-risk prostate cancer. Their cancer must not have spread to other parts of the body.

Design:

The study will last 7 months.

Participants will be screened. They will share their medical history. They will also have:

<TAB>A physical exam

<TAB>Routine blood and urine tests

<TAB>Imaging scans of the chest, abdomen, and pelvis

<TAB>A bone scan

<TAB>A tumor biopsy

<TAB>A specialized MRI. Participants will lie face down on the MRI scanner table. An antenna that receives a signal may be placed in the rectum.

All participants will be treated with radiation therapy and ADT.

Some participants will also receive M9241 as an injection under the skin. This treatment will start 4 weeks after the radiation has ended. Participants will receive a total of 3 doses. The injections will be 4 weeks apart. Some screening tests will be repeated at each visit.

Participants who do not receive M9241 will also have screening tests during the treatment period.

Participants will return for follow-up about 1 month after the last treatment or set of tests.

DETAILED DESCRIPTION:
Background:

* Patients with intermediate and high risk localized prostate cancer often receive radiotherapy with androgen deprivation therapy as a potentially curative treatment. With any local treatment for prostate cancer (radiation or surgery), as many as 20-30% of these intermediate and high risk patients will eventually develop biochemical recurrence within 5 years of treatment.
* There is a growing body of evidence suggesting that stereotactic body radiation therapy (SBRT), which delivers highly conformal high-dose radiation, can promote anti-tumor immune responses both locally and systemically as well as synergize with immune checkpoint inhibitors and other forms of immunotherapy. SBRT is now considered a reasonable alternative to conventional fractionated external beam radiation therapy (EBRT) by the National Comprehensive Cancer Network (NCCN) guidelines and has rapidly proliferated in clinical use.
* M9241 (NHS-IL12) is an immunocytokine composed of two IL-12 heterodimers, each fused to the H-chain of the NHS76 antibody. The NHS76 IgG1 antibody has affinity for both single- and double-stranded DNA (dsDNA) allowing for targeted delivery of proinflammatory cytokine, IL-12, to necrotic portions of tumor at sites of DNA exposure to promote local immunomodulation.
* SBRT-induced dsDNA breaks are tumoricidal and may promote immunogenicity. SBRT also upregulates PD-L1 expression and leads to activation of TGF-Beta. SBRT may enhance intratumoral binding of DNA damage localizing agent, M9241. Preclinical models have demonstrated impressive synergy with radiation plus M9241.
* This study will evaluate the proof of concept that immunocytokines can synergize with standard radiation + ADT in prostate cancer with a focus on T-cell clonality.

Objectives:

* Safety Lead-In: To determine the safety and tolerated doses of the immunocytokine M9241 and Stereotactic Body Radiation Therapy (SBRT) in participants with localized high and intermediate risk prostate cancer receiving standard of care Androgen Deprivation Therapy (ADT)
* To evaluate T-cell clonality, as a measure of immunologic activity, after treatment with SBRT alone or in combination with immunotherapy agent M9241 in participants with prostate cancer receiving standard of care ADT

Eligibility:

* Participants with intermediate or high risk localized prostate cancer
* Participants with no history of prior radiation to the prostate or prior prostatectomy
* Participants without autoimmune disease or history of bleeding disorder
* Participants with adequate organ and bone marrow function

Design:

* This is an open label, randomized, Phase II trial evaluating T-cell clonality after treatment with SBRT alone or in combination with immunotherapy agent M9241in participants with localized intermediate or high risk prostate cancer receiving standard of care ADT.
* The trial will begin with a safety lead-in cohort with de-escalating doses of M9241 (starting dose 16.8 mcg/kg, and de-escalated if needed to 12 mcg/kg, or 8 mcg/kg) only if needed, to evaluate safety and tolerability of the combination of treatments.
* ADT will be administered to all participants on the study as standard care.
* Those participants receiving immunotherapy agents will receive M9241 by subcutaneous injection (sc) at a dose determined during the safety lead-in, every 4 weeks for 3 doses.
* To account for 3 inevaluable participants and 10 screen failures, the accrual ceiling has been set at 65 participants (18 participants during the safety lead-in phase, 34 during the randomized phase II portion).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed localized intermediate or high risk prostate cancer:

  * Intermediate risk - Gleason 7 disease, PSA less than 10
  * High Risk - Gleason 8-10, PSA>10, Extracapsular Extension
* Participants must require treatment with SBRT to the prostate and ADT.
* Pre-treatment tissue availability (collected <= 1 year to initiation of study therapy) for biomarker analysis is mandatory for enrollment. If tissue is determined to be of insufficient/unsuitable quality/quantity, a pre-treatment biopsy prior to initiation of study therapy will be required.
* Male age >= 18 years old
* ECOG performance status < 2
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count >= 1,500/mcL, without CSF support
  * platelets >= 100,000/mcL
  * AST(SGOT)/ALT(SGPT) <= 2.5 X institutional upper limit of normal
  * Hgb >= 10g/dL (pRBC transfusions are not allowed to achieve acceptable Hgb)
  * Total bilirubin <= 1.5 x upper limit of normal (ULN),

OR

in participants with Gilbert s syndrome, a total bilirubin <= 3.0

* Serum albumin >= 2.8 g/dL
* Creatine <= 1.5 X institutional ULN

OR

* Creatinine clearance >= 50 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal by 24h urine
* PT/INR and aPTT <= 1.5 X institutional ULN

  * Testosterone greater than 100 ng/dL.
  * Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) after study entry and for 6 months after completion of radiation treatment or immunotherapy (if taken, whatever is last)
  * Participants must have prostate cancer accessible for biopsy
  * Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Evidence of distant metastatic disease (including clinically or pathologically positive lymph nodes or metastatic disease outside of the pelvis).
* Previous prostatectomy, focal therapy, or radiation to the prostate. Note: Previous finasteride, dutasteride, bicalutamide are allowed at PI discretion.
* Initiation of ADT or SBRT or pelvic nodal radiation irradiation prior to trial enrollment (no time limit).
* Live vaccine therapies for the prevention of infectious disease within 30 days prior to treatment administration. Seasonal flu vaccines that do not contain a live virus are permitted. Locally approved COVID vaccines are permitted.
* Contraindication to mpMRI including allergy or sensitivity to contrast agents (which cannot be alleviated by premedication)
* Contraindications for SBRT such as: rectal wall invasion, history of inflammatory bowel disease, prior radiation in the treatment field that would exceed tissue tolerance.
* Medical comorbidities that preclude the administration of androgen deprivation therapy or uncontrolled chronic or acute intercurrent illness /social situations or other illnesses considered by the Investigator as high risk for investigational drug treatment
* Participants with active immune deficiencies, chronic inflammatory conditions, active autoimmune diseases, or participants on chronic immunosuppressive therapy for whom the primary endpoint of immune response could be impacted.
* Participants requiring requiring systemic corticosteroids (>10 mg daily prednisone equivalent) or immunosuppressive medications except inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Participants with a history of autoimmunity that has not required systemic immunosuppressive therapy or dose not threaten vital organ function including CN, heart, lungs, kidneys, skin and GI track will be allowed
* Participants with HIV
* Active Hepatitis B or Hepatitis C infection
* Significant acute or chronic infections including tuberculosis (history of exposure or history of positive tuberculosis test; plus, presence of clinical symptoms, physical or radiographic findings)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M9241.
* Participants with prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast or low risk Gleason 6 prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine safety and tolerated doses of M9241 and SBRT | four weeks after start of treatment
  For the safety lead-in: grade and type of toxicities at each dose level will be assessed to determine safety and tolerated doses of M9241 in combination with SBRT in participants with high and intermediate risk prostate cancer receiving standard of care ADT
evaluate T-cell clonality as measures of immunologic activity | baseline through 4 weeks after end of treatment
  Relative T-cell antigen receptor (TCR) clonality for each participant will be formed and these ratios will be compared between the two arms.

SECONDARY OUTCOMES:
Evaluate peripheral immune response | baseline through 4 weeks after end of treatment
  Immune cell subsets will be evaluated to determine peripheral immune response and compare between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing will be shared with subscribers to dbGAP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as the database is active
Access Criteria: Clinical data will be made available via subscription to BTRIS and with permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000114-C.html